CLINICAL TRIAL: NCT04397874
Title: Maternal Perception of Fetal Movements Evaluation Using and Analyzing the Variables of Antepartum Computerized Cardiotocography: An Exploratory Study.
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, MD, research , gynecology and obstetrics, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 003
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Fetal Movement
Keywords: Fetal movement; Fetal activity; fetal assessment; fetal well-being; Computerized cardiotocography (cCTG); Fetal heart rate (FHR)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ; Computerized cardiotocography (cCTG) — To estimate the correlation between the maternal perception of fetal movement and antepartum computerised cardiotocography parameters.

SUMMARY:
Several studies analysed the association of fetal movement counting with perinatal mortality and fetal outcomes. However, no one examined the relationship of the maternal perception of fetal movement with the fetal wellbeing quantifies through computerised cardiotocography.

Our study evaluates the correlation between the maternal perception of fetal movement and antepartum computerised cardiotocography parameters.

ELIGIBILITY:
Inclusion Criteria:

* nonlaboring term singleton pregnancies (37 0/7 - 41 6/7 weeks of gestation)

Exclusion Criteria:

* fetal malformations, stillbirths, preterm deliveries

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: physiological nonlaboring term singleton pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To estimate the correlation between the maternal perception of fetal movement and antepartum computerised cardiotocography parameters. | External cCTG was completed at least 20 minutes (maximum 60 minutes), two transducers were placed on the maternal abdomen: one over the fetal heart level and the other one at the uterine fundus. For each cCTG, the following data were evaluated: Basal FHR

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi della Campania "Luigi Vanvitelli"- OB & Gyn -, Napoli, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided